CLINICAL TRIAL: NCT02517073
Title: A Survey on the Practice of Mechanical Ventilation Among Patients With Severe Brain Injury in China: a Prospective Observational Study
Brief Title: Practice of Mechanical Ventilation in Patients With Severe Brain Injury in China
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: MCS-2015-008
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Respiration, Artificial
Keywords: mechanical ventilation; epidemiology; intensive care unit; national survey
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The mechanical ventilation strategy has changed over years worldwide. Several international researches have been conducted to study the association of the use of mechanical ventilation with clinical outcomes. In this prospective, multicenter, cross-sectional survey, the practice of mechanical ventilation among patients with severe brain injury will be investigated in 70 intensive care units in China.

ELIGIBILITY:
Inclusion Criteria:

1. older than 18 years
2. with severe brain injury (including severe traumatic brain injury, ischemic stroke, subarachnoid hemorrhage, spontaneous intracerebral hemorrhage, hypoxic-ischemic encephalopathy, intracranial tumor, intracranial infection and idiopathic epilepsy)
3. mechanical ventilated for at least 24 hours before the time of on-spot survey

Exclusion Criteria:

1. undergoing a spontaneous breathing trial (SBT) at the time of on-spot survey
2. underwent at least once SBT in the preceding 24 hours before time of on-spot survey
3. enrolled in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanical ventilated patients with severe brain injury
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of patients receiving control and assist mode of mechanical ventilation | During 1 hour of on-spot survey
  Control mode is defined as volume or pressure control ventilation. Assist mode is defined as synchronized intermittent mandatory ventilation and pressure support ventilation.

SECONDARY OUTCOMES:
The settings of tidal volume, inspiratory pressure, and positive end-expiratory pressure in enrolled patients | During 1 hour of on-spot survey
Duration of mechanical ventilation | 60 days after on-spot survey
Number of patients liberated from mechanical ventilation | 60 days after on-spot survey
Neurological outcome by Glasgow Outcome Scale | 60 days after on-spot survey

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — Acute Brain Injury and Critical Care Research Collaboration, ABC Research Collaboration
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Luo XY, Hu YH, Cao XY, Kang Y, Liu LP, Wang SH, Yu RG, Yu XY, Zhang X, Li BS, Ma ZX, Weng YB, Zhang H, Chen DC, Chen W, Chen WJ, Chen XM, Du B, Duan ML, Hu J, Huang YF, Jia GJ, Li LH, Liang YM, Qin BY, Wang XD, Xiong J, Yan LM, Yang ZP, Dong CM, Wang DX, Zhan QY, Fu SL, Zhao L, Huang QB, Xie YG, Huang XB, Zhang GB, Xu WB, Xu Y, Liu YL, Zhao HL, Sun RQ, Sun M, Cheng QH, Qu X, Yang XF, Xu M, Shi ZH, Chen H, He X, Yang YL, Chen GQ, Sun XM, Zhou JX; Acute Brain Injury and Critical Care Research Collaboration (ABC Research Collaboration). Lung-protective Ventilation in Patients with Brain Injury: A Multicenter Cross-sectional Study and Questionnaire Survey in China. Chin Med J (Engl). 2016 Jul 20;129(14):1643-51. doi: 10.4103/0366-6999.185869. PMID 27411450